CLINICAL TRIAL: NCT02097602
Title: Can Reticulated Platelets Predict the Outcome After Noncardiac Surgery?
Brief Title: Correlation Between Reticulated Platelets and Major Adverse Cardiac and Cerebrovascular Events After Noncardiac Surgery
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: RePOS
Record Dates: First submitted 2014-03-17; First posted 2014-03-27 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Cardiac Death; Congestive Heart Failure; Angina Pectoris; Stroke; Pulmonary Embolism; Deep Vein Thrombosis
Keywords: Reticulated platelets; noncardiac surgery; MACCEs; major adverse cardiac and cerebrovascular events; outcome; High-risk or intermediate-risk noncardiac surgery
MeSH Terms: conditions — Death; Heart Failure; Angina Pectoris; Stroke; Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is an observational study designed to monitor the course of the fraction of reticulated platelets and the correlation thereof to major adverse cardiac and cerebrovascular events after noncardiac surgery.

DETAILED DESCRIPTION:
Reticulated platelets (RP) are newly formed, immature platelets which in contrast to mature platelets have high granule content and a residual amount of mRNA. An increased mean platelet volume (MPV) and the fraction of RP have been shown to be correlated to cardiovascular events like myocardial infarction or cardiovascular death. However, there are no trials so far investigating how surgery impacts the fraction of RP and how this fraction correlates with the outcome after noncardiac surgery.

Patients with an age above 18 years undergoing high-risk or intermediate-risk noncardiac surgery are to be included. The fraction of RP is to be investigated in routinely acquired blood samples preoperatively, postoperatively in the recovery room, as well as 24-72 hours after anaesthesia and surgery.

A primary common endpoint are major adverse cardiac and cerebrovascular events (MACCEs), as well as deep vein thrombosis and pulmonary embolism. MACCEs are defined according to Sabaté et al. as: cardiac death, cerebrovascular death, nonfatal cardiac arrest, acute myocardial infarction, congestive heart failure, new cardiac arrhythmia, angina or stroke. Secondary endpoints are lengths of hospital stay and intensive care stay as well as mortality after 3 months. All participants are to be contacted by phone three months after discharge and their health situation is to be determined.

1000 patients will be enrolled in a defined time frame of six months

ELIGIBILITY:
Inclusion Criteria:

* high-risk or intermediate-risk surgical patients undergoing noncardiac surgery
* age ≥ 18 years
* written informed consent

Exclusion Criteria:

* low-risk surgery
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High-risk or intermediate-risk surgical patients older than 18 years undergoing noncardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
major adverse cardiac and cerebrovascular events (MACCEs) | during the hospital stay, an expected average of 2 weeks
  MACCEs are defined according to Sabaté et al. as: cardiac death, cerebrovascular death, nonfatal cardiac arrest, acute myocardial infarction, congestive heart failure, new cardiac arrhythmia, angina or stroke. Pulmonary embolism and deep vein thrombosis are further primary endpoints.

SECONDARY OUTCOMES:
Mortality | three months after discharge
  mortality
length of hospital and intensive care-stay | three months after discharge
  length of hospital and intensive care-stay

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Jungwirth, MD, Study Director — Klinikum rechts der Isar Technische Universität München; Aida Anetsberger, MD, Principal Investigator — Klinikum rechts der Isar Technische Universität München
Locations (1):
- Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München, Ismaninger Str. 22, Munich, Germany

REFERENCES:
- [Background] Nakamura T, Uchiyama S, Yamazaki M, Okubo K, Takakuwa Y, Iwata M. Flow cytometric analysis of reticulated platelets in patients with ischemic stroke. Thromb Res. 2002 May 15;106(4-5):171-7. doi: 10.1016/s0049-3848(02)00131-7. PMID 12297121
- [Background] Grove EL, Hvas AM, Kristensen SD. Immature platelets in patients with acute coronary syndromes. Thromb Haemost. 2009 Jan;101(1):151-6. PMID 19132202
- [Background] Cesari F, Marcucci R, Gori AM, Caporale R, Fanelli A, Casola G, Balzi D, Barchielli A, Valente S, Giglioli C, Gensini GF, Abbate R. Reticulated platelets predict cardiovascular death in acute coronary syndrome patients. Insights from the AMI-Florence 2 Study. Thromb Haemost. 2013 May;109(5):846-53. doi: 10.1160/TH12-09-0709. Epub 2013 Mar 14. PMID 23494003
- [Background] Sabate S, Mases A, Guilera N, Canet J, Castillo J, Orrego C, Sabate A, Fita G, Parramon F, Paniagua P, Rodriguez A, Sabate M; ANESCARDIOCAT Group. Incidence and predictors of major perioperative adverse cardiac and cerebrovascular events in non-cardiac surgery. Br J Anaesth. 2011 Dec;107(6):879-90. doi: 10.1093/bja/aer268. Epub 2011 Sep 2. PMID 21890661
- [Derived] Anetsberger A, Bernlochner I, Jungwirth B, Blobner M, Meyer B, Kochs EF, Bongiovanni D, Schmid S, Langgartner C, Baumgart L, Gempt J. Association of immature platelets with perioperative complications in neurosurgery. Platelets. 2023 Dec;34(1):2185462. doi: 10.1080/09537104.2023.2185462. PMID 36974887
- [Derived] Anetsberger A, Blobner M, Haller B, Schmid S, Umgelter K, Hager T, Langgartner C, Kochs EF, Laugwitz KL, Jungwirth B, Bernlochner I. Immature platelets as a novel biomarker for adverse cardiovascular events in patients after non-cardiac surgery. Thromb Haemost. 2017 Oct 5;117(10):1887-1895. doi: 10.1160/TH16-10-0804. Epub 2017 Aug 10. PMID 28796275